CLINICAL TRIAL: NCT06018389
Title: Prevention of Hazardous Use of Alcohol Among High School Students in Denmark: a Cluster Randomized Controlled Trial
Brief Title: Prevention of Hazardous Use of Alcohol with Danish High School Students (Our Choice)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: voresvalg_40833; 2022-0367531 seqno. 3073 (Other: AU record, University of Aarhus); ID: 155933 (Other: TrygFonden)
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Healthy Participants
Keywords: Prevention; High School; Alcohol; Substance Use; Adolescents; Motivational Interviewing; School Policies; Parents
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The study employs a parallel group cluster randomized controlled trial design with three conditions: 1) structural condition targeting school and parent levels, 2) structural condition combined with group MI which also targets the student level, and 3) assessment-only control condition (interventions offered after the last follow-up survey).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Structural Only (Experimental): The Structural Only condition consists of (1) school policies for school-based social events; and (2) an information-based interactive parent meeting. Interventions in this arm are targeting the school and parent level.
  Interventions: Behavioral: Structural only
- Structural+Group MI (Experimental): The Structural+Group MI condition consists of the elements described in "Structural Only" and group MI. Interventions in this arm are targeting all three levels: school, parent and student level.
  Interventions: Behavioral: Structural only; Behavioral: Structural+Group MI
- Control (No Intervention): The Control condition is an assessment-only condition. During the period under study, it includes the same assessments (surveys) as the other two conditions. After the last follow-up (August 2024), control schools can opt-in to receive any of the intervention programs.

INTERVENTIONS:
Behavioral: Structural only — A shared list of school policies for or related to, school-based social events at school premises. The policy initiatives include (but are not limited to): increasing the number of social events without alcohol; promoting non-alcoholic beverages at parties; working with student associations regarding their roles and responsibilities; encouraging parental involvement at school events and disseminating the schools' alcohol policy among students and parents. The school principal and management will be responsible for the implementation and enforcement of the policies.
  The Information-based interactive parent meetings will be 45 minutes and will take place at the schools. Parents will be offered concrete, research-informed advice about how they can reduce risk of hazardous substance use and promote well-being among their adolescents. Following a 15-minute presentation, the group leader facilitates a discussion and exchange of experience between parents.
  Arms: Structural Only; Structural+Group MI
Behavioral: Structural+Group MI — Within school classes, students are divided into groups of 5-8 students and each group will be assigned a group leader from the research team. The group-based Motivational Interviewing (group MI) is manualized and consists of two one-hour group sessions administered over two consecutive weeks. The first session is focused on "Tell your story", "Gains from not drinking", and "Social norms." In the second session, the focus is on "Personal values", "Linking values with behavior" and "Planning/choices regarding alcohol". Both group MI sessions will take place at the schools during the school day.
  Arms: Structural+Group MI

SUMMARY:
The trial 'Our Choice' examines the effect of two prevention interventions targeting school, parent, and student levels at Danish high schools. The interventions aim to reduce hazardous use of alcohol and related health outcomes among first-year students in Denmark (ages 15-18). The investigators hypothesizes that a structural intervention (school and parent levels) reduces hazardous alcohol use and related health outcomes compared to an assessment-only control group 12 months post baseline; and that adding group-based Motivational Interviewing (group MI) yields further improvements. Additionally, factors related to the implementation of the interventions are examined.

DETAILED DESCRIPTION:
The main aim of the 'Our Choice' cluster randomized controlled multisite trial is to test the efficacy of interventions aimed at reducing hazardous use of alcohol and related health outcomes among first-year students (15-18 years) in high schools in Denmark. Furthermore, the aim is to examine feasibility and acceptability of the interventions with Danish students in high school, as well as with staff (e.g., teachers and principals) to inform future implementation studies.

The study employs a parallel group cluster randomized controlled trial design with three conditions:

1. Structural condition targeting school and parent levels via school policies for school-based social events and an information-based interactive parent meeting.
2. Structural condition combined with group-based Motivational Interviewing (group MI) which also targets the student level.
3. Assessment-only control condition with the same assessments as the other two conditions and with interventions offered after the last follow-up survey.

The study hypothesizes that students in the structural condition (school and parent levels) reduce hazardous alcohol use and related health outcomes compared to students in the assessment-only control condition 12 months post baseline; and that adding group MI yields further improvements.

A participatory approach is used to adapt and develop interventions. Sixteen high schools in Denmark and N=3100 first-year students enrolled in high school in August 2023 will be recruited. Data will be collected via online questionnaires pre-interventions (baseline), 2, 6, 9 and 12 months post baseline. The primary outcome will be analyzed with generalized linear mixed models. Feasibility and acceptability will be assessed via surveys (students) and interviews (high school staff) to inform future implementation.

ELIGIBILITY:
Inclusion Criteria:

* Students starting high school in one of the 16 participating high schools in August 2023
* Minimum 15 years old
* Understand and speak Danish
* Able to give independent informed consent
* Staff (school principals, teachers, or administrative employees) from one of the 16 participating high schools

Exclusion Criteria:

* Under 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3100 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Past month high-intensity drinking | From baseline to 12 months after baseline
  Past month high-intensity drinking: peak drinks per drinking event, assessed with the Timeline FollowBack (TLFB) (count measure)

SECONDARY OUTCOMES:
Past month alcohol-related consequences | From baseline to 12 months after baseline
  Assessed by 21 items covering physical, social and mental issues related to hazardous use of alcohol, developed by the team for Danish youth based on single items from previous Danish surveys and the Rutgers Alcohol Problems Index e.g. black-outs, (emotional) hangovers), sexual contact that was later regretted, with yes/no response options (summed score: range 0-21) with higher scores indicating more negative consequences.
Past month heavy episodic drinking events | From baseline to 12 months after baseline
  Past month heavy episodic drinking events assessed by TLFB (count measure).
Well-being in class | From baseline to 12 months after baseline
  Assessed by six items rated on a five-point scale from 'completely disagree' to 'completely agree' e.g., I feel accepted by the others in my class (summed score: range 0-30) with a score of 30 representing the best possible well-being in class.
World Health Organization Five Well-being Index (WHO-5) | From baseline to 12 months after baseline
  Psychological well-being, assessed by The World Health Organization Five Well-being Index (summed score: range 0-25) with a score of 25 representing the best possible quality of life.
Past month use of tobacco | From baseline to 12 months after baseline
  Measured by days using tobacco (count measure: range 0-30 days)
Past month use of illegal substances | From baseline to 12 months after baseline
  Measured by days using cannabis, cocaine, and other illegal drugs (count measure: range 0-30 days).

CONTACTS AND LOCATIONS:
Overall Officials: Krisrtine Rømer Thomsen, Principal Investigator — Centre for Alcohol and Drug Research, Aarhus BSS, Aarhus University
Locations (1):
- Centre for Alcohol and Drug Research, Aarhus BSS, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
After the conclusion of the study, data from the study will be made available by the Centre for Alcohol and Drug Research, Aarhus University, upon reasonable request, and within the limitations set by the Danish data protection legislation and regulation.

REFERENCES:
- [Background] Romer Thomsen K, Vallentin-Holbech L, Xylander S, Wellnitz KB, Tolstrup J, Nielsen AS, Ewing SWF. Prevention of hazardous use of alcohol among high school students: a study protocol for the randomized controlled trial 'Our choice'. BMC Public Health. 2023 Oct 24;23(1):2079. doi: 10.1186/s12889-023-16976-y. PMID 37875851